CLINICAL TRIAL: NCT06324643
Title: Effect of Sensory Motor Training on Activities of Daily Living in Erb's Palsy Childern
Brief Title: Sensory Motor Integration Training in Erb's Palsy Childern
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sara Elsayed Ali Abdelnaby Ali (Other)
Responsible Party: Sponsor-Investigator, Sara Elsayed Ali Abdelnaby Ali, sara elsayed ali abdelnaby, Kafrelsheikh University
Organization: Kafrelsheikh University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Erb's Palsy
Record Dates: First submitted 2024-03-15; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Sensory Motor Integration and Erb's
Keywords: Erb's palsy -sensory motor integration - ADL- Bimanual hand use

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Use Designed occupational therapy program in childern with erb's palsy (Experimental): 1st group treated by strengthening exercises , stretching ,and occupational therapy
  Interventions: Procedure: sensory motor integration training
- Use designed occupational therapy program and sensory motor integration training (Experimental): 2nd group treated by strengthening exercises , stretching ,and occupational therapy and sensory motor integration training (use different textures and different temperature)
  Interventions: Procedure: sensory motor integration training

INTERVENTIONS:
Procedure: sensory motor integration training — one group treated by strengthening exercises , stretching ,and occupational therapy and other group treated by strengthening exercises , stretching ,and occupational therapy and sensory motor integration training

SUMMARY:
The aim of the study is to Study effect of sensory motor integration training on ADL activities in children with Erb's palsy.

DETAILED DESCRIPTION:
Thirty-two participants , their age ranged from two to six years for both genders (sixteen children treated with designed occupational therapy program group A and sixteen treated with designed occupational therapy program and sensory motor integration training group B )

ELIGIBILITY:
Inclusion Criteria:

1. Their ages will be ranged from 2 to 6 years in both sexes.
2. The infants with Erb's palsy (C5-C6).
3. Can follow verbal commend
4. Muscle tone within normal and muscle power within functional range.
5. Intact vision and hearing.

Exclusion Criteria:

1. Children undergoing surgical treatment.
2. Cognitive problem and cognitive anomalies.
3. Children with Erb's engram.
4. Complete sensory loss.
5. Shoulder subluxation or dislocation.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 35 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Effect of sensory motor integration training on ADL | 3 months
  Assessment of bimanual performance and family-reported upper-extremity use by Assisting Hand Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Sara Elsayed ali abdelnaby, Bachelor's, Principal Investigator — Kafrelsheikh University; Abd Elaziz Ali sherif, Study Chair — Professor of pediatric department- Faculty of physical therapy- kafrelsheikh university; Osama Abd Elfattah El-Agamy, Study Chair — professor and head of department of pedateric-faculty of medicine -kafrelsheik university; Sara Yousef Abdel Elglil Elsebahy, Study Director — Lecturer of pediatric department -Faculty of physical therapy- Kafrelshiekh University